CLINICAL TRIAL: NCT05239585
Title: Pilot Study on the Use of a Wearable Remote Electroencephalography Device to Identify Neonates at Risk for Neonatal Seizures and Status Epilepticus
Brief Title: Remote EEG Device for Identification of Risk for Neonatal Seizures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to finalize technology for use in study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anthony L. Fine, MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 21-006001
Record Dates: First submitted 2022-01-05; First posted 2022-02-15 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Remote EEG monitoring (Experimental): All subjects will pilot the use of wireless EEG technology in neonates with mild neonatal encephalopathy and neonates with spells to see if this device can be used to determine the risk for neonatal seizure and need for escalation of care and full scalp EEG
  Interventions: Device: Epilog device

INTERVENTIONS:
Device: Epilog device — Pilot the use of wireless EEG technology in neonates with mild neonatal encephalopathy and neonates with spells to see if this device can be used to determine the risk for neonatal seizure and need for escalation of care and full scalp EEG

SUMMARY:
The purpose of this study is to see if the use of wireless brain wave monitoring can be helpful for newborns and help their medical providers identify seizures earlier and to monitor for the risk for seizures.

DETAILED DESCRIPTION:
Our goals are to evaluate the effectiveness of the Epilog device in identification of neonates who are at risk for seizures and need formal EEG monitoring or cooling. The current process for these patients would be transfer from Rochester Methodist Hospital to the St. Mary's level 3 NICU for EEG monitoring. Given that in case of neonatal encephalopathy, there is 6-hour window in which to make the critical decision of whether to initiate therapeutic hypothermia or not, rapid access to EEG data is crucial. We would like to perform a pilot study on use of wireless EEG technology in neonates with mild neonatal encephalopathy and neonates with spells to see if this device can be used to determine the risk for neonatal seizure and need for escalation of care and full scalp EEG.

ELIGIBILITY:
Inclusion Criteria:

* Age 28 days old or less (postnatal age)
* Neonatal encephalopathy as judged by clinical team or symptoms concerning for subtle seizures
* Patient currently in level 1 newborn nursery or level 2 or 3 NICU

Exclusion Criteria:

* Medical comorbidity which would result in prolonged need for sedation
* Prolonged EEG monitoring is medically indicated

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the Epilog device in identification of neonates who are at risk for seizures and need formal EEG monitoring or cooling | Approximately 2 to 72 hours
  Total number of neonates that Epilog device identifies as requiring formal EEG monitoring
Evaluate time to formal long-term EEG monitoring in neonates monitored with the Epilog device compared to a historical control cohort of neonates undergoing EEG evaluation. | Approximately 2 to 72 hours
  Time from initiation of monitoring with Epilog device to monitoring completion or conversion to formal prolonged EEG monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony L Fine, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States